CLINICAL TRIAL: NCT00392509
Title: A Phase I-II Randomized Autologous Bone Marrow Derived Aldehyde Dehydrogenase-Bright (ALDHbr) Cells Against Unfractionated Autologous Mononuclear Bone Marrow in Patients With Rutherford 4 or 5 Peripheral Arterial Occlusive Disease
Brief Title: ALD-301 for Critical Limb Ischemia, Randomized Trial
Acronym: CLI-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aldagen (Industry)
Responsible Party: Laurence Keller, MD, Aldagen, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BB IND 12875
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease; Peripheral Vascular Disease
Keywords: critical limb ischemia; cell therapy for angiogenesis; aldehyde dehydrogenase-bright cells; peripheral artery disease; peripheral vascular disease; leg pain; PVD; PAD; CLI; amputation; limb salvage
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Experimental): Unfractionated Autologous Mononuclear Bone Marrow
  Interventions: Procedure: ALDH-br bone marrow cells vs. mononuclear bone marrow cells

INTERVENTIONS:
Procedure: ALDH-br bone marrow cells vs. mononuclear bone marrow cells — Surgery

SUMMARY:
This study will treat patients with such severe lower leg ischemia or vascular compromise that they have pain at rest. The goal is to compare treatment of the patient's painful disorder by injecting cells into the calf of the leg and testing for circulatory improvement. A treatment will given at random to two groups and will be injection into the calf muscle with ALD-301 (specially processed stem and progenitor cells) from the patient's own bone marrow, or with cells processed by more routine that minimally purifies the cells. The study goal is to see if the ALD-301 cells are more effective in generating new small blood vessels to improve the circulation to the affected leg.

DETAILED DESCRIPTION:
Patients will be recruited who have critical limb ischemia with pain at rest. The study will select patients for treatment and follow them for three months after intervention. The treatment will consist of drawing about 2/3 of a cup of bone marrow from the patient's hip bone, then processing the collected bone marrow will be as follows:

* The test group's bone marrow will be processed and sorted to identify the aldehyde dehydrogenase bright ALDH-br stem and progenitor cells (ALD-301). These cells will be injected into the calf muscle of the patient in clinic.
* The control group will have the same amount of bone marrow collected but it will undergo a simpler process to isolate the mononuclear cells from the whole bone marrow, removing most of the red cells and granulocytes from cell preparation for injection.

The patients will be monitored for adverse events related to this process to determine the safety of the approach. They will also be tested at intervals during the study to compare baseline values of each patient with the post-treatment values of:

1. ankle-brachial index of systolic blood pressure
2. the transcutaneous oxygen measurements obtained from the skin of the treated leg
3. the patient's perception of his/her quality of life as measured by two different, validated questionnaires
4. Measurements of of heel/foot ulcers, if present, to monitor degree of healing if it occurs
5. the patient's perception of his/her level of pain in the leg

The patients will receive a call at 6 months to report on additional life events following the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or greater with atherosclerotic vascular disease that is viewed as not readily amenable to reconstructive surgery and Rutherford Category 4 ischemia (ischemic rest pain) and Rutherford Category 5 ischemia (ulceration or tissue necrosis) and by the judgment of their referring physician are not reasonable candidates for revascularization options of either percutaneous balloon angioplasty or a surgical revascularization.
* Objective evidence of severe peripheral arterial disease will include an ankle brachial index (ABI) of less than 0.5, or, in the case of patients who have vessels calcified and thereby "non-compressible" vessels metatarsal pulse volume recording (PVR) that is flat or barely pulsatile in the diseased limb on two consecutive examinations performed at least one week apart.
* Patients competent to give informed consent.
* No active malignant disease that could involve the bone marrow, or history of treatment of malignant disease that could have damaged the bone marrow.
* Before being accepted for the study the patient must be screened for human immunodeficiency virus, hepatitis B virus, hepatitis C virus, human transmissible spongiform encephalopathy, including Creutzfeldt-Jacob Disease, Treponema pallidum, and have a negative standard infectious disease panel including a CMV PCR test.
* Patients who are hemodynamically stable.

Exclusion Criteria:

* Patients with poorly controlled diabetes mellitus (HbA1C > 8%)
* Patients with renal insufficiency (creatinine > 2.5).
* Patients with evidence of infectious disease as determined by e. above or other medical findings.
* Pregnant women (women capable of childbearing must have a negative pregnancy test).
* Patients with cognitive impairments.
* Other comorbid disease that would be expected to result in less than one year life expectancy
* Past malignancy or history of chemotherapy or radiation affecting the bone marrow.
* History of inflammatory or progressively fibrotic conditions: .e.g., rheumatoid arthritis, systemic lupus erythematosis, vasculitic disorders, idiopathic pulmonary fibrosis, retroperitoneal fibrosis
* Infection as evidenced by WBC count of >15,000 and/or temperature >38 degrees C. Large area of cellulitis in the afflicted limb that in the opinion of the investigators would require the institution of antibiotics OR evidence of osteomyelitis corroborated by radiographic or scintigraphic examination
* Cardiovascular conditions:

  * Exercise limiting angina ( Canadian Cardiovascular Society Class 3 (Appendix 7);
  * Congestive heart failure (New York Heart Association class 3 (Appendix 5);
  * Unstable angina;
  * Acute ST elevation myocardial infarction (MI) within 1month;
  * Transient ischemic attack or stroke within 1 month;
  * Severe valvular disease
* Patients with any history of organ transplants;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
adverse events | 6 months
ankle-brachial systolic pressure index | 3 mo
transcutaneous oxygen value (mm Torr) | 3 mo
quality of life (questionnaires) | 3 mo

SECONDARY OUTCOMES:
size of lower extremity ulcer(s) | 3 mo
peripheral nerve conduction exam | 3 mo
level of pain at rest (questionnaire) | 3 mo
limb clinical status | 3 mo

CONTACTS AND LOCATIONS:
Overall Officials: Emerson C Perin, M.D., Ph.D., Principal Investigator — Stem Cell Center, Texas Heart Institute, St Luke's Episcopal Hospital, 6770 Bertner , Suite 1020 Texas Medical Center,Houston, Texas 77030; Robert Mitchell, MD, Principal Investigator — Duke University; Michael Murphy, MD, Principal Investigator — University of Indiana at Indianapolis; Nicolas Chronos, MD, Principal Investigator — Saint Joseph's Research Institute; Farrell Mendelsohn, MD, Principal Investigator — Cardiology PC
Locations (5):
- United States (5):
  - Cardiology PC, Birmingham, Alabama
  - Saint Joseph's Research Institute, Atlanta, Georgia
  - University of Indiana at Indianapolis, Indianapolis, Indiana
  - Duke University Medical Center, Durham, North Carolina
  - Texas Heart Institute, Stem Cell Center, 6770 Bertner, St Luke's Episcopal Hospital, Houston, Texas

REFERENCES:
- [Derived] Perin EC, Silva G, Gahremanpour A, Canales J, Zheng Y, Cabreira-Hansen MG, Mendelsohn F, Chronos N, Haley R, Willerson JT, Annex BH. A randomized, controlled study of autologous therapy with bone marrow-derived aldehyde dehydrogenase bright cells in patients with critical limb ischemia. Catheter Cardiovasc Interv. 2011 Dec 1;78(7):1060-7. doi: 10.1002/ccd.23066. Epub 2011 May 18. PMID 21594960
- See also: Sponsor's Website — http://www.aldagen.com